CLINICAL TRIAL: NCT03417089
Title: Suspension of Falciform Ligament During Mini Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fac.med.052
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Upper GIT Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- falciform ligament suspension (Experimental): routine suspension of falciform ligament during mini gastric bypass,
  Interventions: Procedure: Falciform ligament suspension
- No suspension (Active Comparator): working without suspension of the falciform ligament
  Interventions: Procedure: no suspension

INTERVENTIONS:
Procedure: Falciform ligament suspension — routine of falciform ligament suspension during Mini gastric bypass
  Arms: falciform ligament suspension
Procedure: no suspension — working without of falciform ligament suspension during Mini gastric bypass
  Arms: No suspension

SUMMARY:
The falciform ligament is hanging down in the upper abdomen and usually impede the work during laparoscopic upper GIT surgery, especially in obese patient, so the aim of this study is to evaluate the impact of routine suspension of falciform ligament during mini gastric bypass, which is advanced laparoscopic procedure, by comparing the outcomes in 2 groups of patient in the fist group the investigators will routinely suspend the falciform ligament and the other group the investigators will working without suspension

DETAILED DESCRIPTION:
The falciform ligament is hanging down in the upper abdomen and usually impede the work during laparoscopic upper GIT surgery, especially in obese patient, so the aim of this study is to evaluate the impact of routine suspension of falciform ligament during mini gastric bypass, which is advanced laparoscopic procedure, by comparing the outcomes in 2 groups of patient in the fist group the investigators will routinely suspend the falciform ligament and the other group the investigators will working without suspension

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patient with BMI more than 40 with or without co-morbidity
* Morbidly obese patient with BMI more than 35 with co-morbidity

Exclusion Criteria:

* Unfit patients for laparoscopic sleeve gastrectomy
* Patients refuse to share in the study
* Patients that already on PPI due to any indications
* Revisional surgery for obesity
* Previous upper abdominal surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
the difficulty of working during mini gastric bypass | 5 hours
  difficulty of working during mini gastric bypass assessed by many parameters like number of clashing of instruments per one operations and operative time

SECONDARY OUTCOMES:
operative time | 6 hours
  duration of the operation from skin to skin

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Sewefy, MD, Principal Investigator — Minia University
Locations (1):
- Faculty of medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided